CLINICAL TRIAL: NCT02926885
Title: Efficacy Evaluation of the Esophagogastric Junction Exposure Obtained by the Flexible Liver Retractor in Gastroplasty for Obesity
Brief Title: Efficacy Evaluation of the Esophagogastric Junction Exposure Obtained by the Flexible Liver Retractor in Gastroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara (Other)
Responsible Party: Principal Investigator, RODRIGO FEITOSA DE ALBUQUERQUE LIMA BABADOPULOS, MD, GASTRIC SURGEON, Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RB001
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
Keywords: liver; laparoscopy; Bariatric Surgery; Esophagogastric Junction; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONVENTIONAL LIVER RETRACTOR DEVICE (Active Comparator): USE OF CONVENTIONAL LIVER RETRACTOR FOR THE LAPAROSCOPIC ROUX-EN-Y GASTRIC BYPASS SURGERY
  Interventions: Device: CONVENTIONAL LIVER RETRACTOR DEVICE; Procedure: LAPAROSCOPIC ROUX-EN-Y GASTRIC BYPASS SURGERY
- FLEXIBLE LIVER RETRACTOR DEVICE (Experimental): USE OF THE FLEXIBLE LIVER RETRACTOR FOR THE LAPAROSCOPIC ROUX-EN-Y GASTRIC BYPASS SURGERY
  Interventions: Device: FLEXIBLE LIVER RETRACTOR DEVICE; Procedure: LAPAROSCOPIC ROUX-EN-Y GASTRIC BYPASS SURGERY

INTERVENTIONS:
Device: CONVENTIONAL LIVER RETRACTOR DEVICE — LIVER RETRACTION FOR THE EXPOSURE OF THE ESOPHAGOGASTRIC JUNCTION USING CONVENTIONAL RETRACTOR DEVICE
  Arms: CONVENTIONAL LIVER RETRACTOR DEVICE
Device: FLEXIBLE LIVER RETRACTOR DEVICE — LIVER RETRACTION FOR THE EXPOSURE OF THE ESOPHAGOGASTRIC JUNCTION USING FLEXIBLE LIVER RETRACTOR DEVICE
  Arms: FLEXIBLE LIVER RETRACTOR DEVICE
Procedure: LAPAROSCOPIC ROUX-EN-Y GASTRIC BYPASS SURGERY — LAPAROSCOPIC ROUX-EN-Y GASTRIC BYPASS SURGERY

SUMMARY:
Evaluation of a new technique of liver retraction for the exposure of the His angle in gastric bypass Roux-en-Y surgery.

DETAILED DESCRIPTION:
Obesity is a chronic disease of clinical treatment initially, but with precise surgical indications regulated by national and international health organizations. Among the surgical techniques, the gastric bypass Roux-en-Y is considered the "gold standard" for its efficiency and low morbidity and mortality. In gastric laparoscopic surgery it is necessary to move the liver in order to ensure adequate working space and a good view. Conventional laparoscopic retractors surgery are generally coarse, require an additional incision for its installation, or handling by an assistant during surgery and involve risk of liver injury. The objective of this study was to evaluate the efficacy of a flexible liver retractor in the exposure of the His angle in Roux-en-Y gastric bypass for morbid obesity. This was a prospective, controlled, open and comparative study, with 100 patients randomly divided into two groups (conventional and flexible retractor), with medical indication for bariatric surgery. Data were recorded during surgery in both groups for comparison of the two hepatic retraction techniques.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 - 65 years, both genders, with indication of bariatric surgery according to IFSO criteria.
* Agreed to participate and signed informed consent form.

Exclusion Criteria:

* Patients who did not agree to participate and / or any other condition that the investigator judged relevant for not participating in the study were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of incisions made during laparoscopic surgery using flexible retractor when compared to conventional retractor | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Babadopulos, MD, Principal Investigator — Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara
Locations (1):
- Nucleo de Pesquisa e Desenvolvimento da Universidade Federal do Ceara, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No